CLINICAL TRIAL: NCT03328325
Title: Evaluation of the Effects of Age, Prior Exposure, and Previous Vaccination on the B Cell Response to Inactivated Influenza Vaccine in Healthy Adults and Children
Brief Title: Age and Response to Flu Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-0101; HHSN272201400005C; NCT03133936 (obsolete NCT alias)
Record Dates: First submitted 2017-10-26; First posted 2017-11-01 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-03-03

CONDITIONS: Influenza; Influenza Immunisation
Keywords: B Cell Response; Children; Evaluation; Healthy Adults; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): 0.5 mL dose of quadrivalent (IIV-4) vaccine administered once intramuscularly, n=240
  Interventions: Biological: Influenza Virus Quadrivalent Inactivated Vaccine

INTERVENTIONS:
Biological: Influenza Virus Quadrivalent Inactivated Vaccine — A seasonal quadrivalent inactivated influenza vaccine (IIV4), prepared from influenza viruses propagated in embryonated chicken eggs, protecting against 2 influenza A subtypes and 2 influenza B subtypes: A/Singapore/GP1908/2015 (H1N1) IVR-180 (an A/Michigan/45/2015 [H1N1] pdm09-like virus), A/Singapore/INFIMH-16-0019/2016 (H3N2) IVR-186, B/Maryland/15/2016 NYMC BX-69A, (a B/Colorado/06/2017-like virus), and B/Phuket/3073/2013.
Biological: Influenza Virus Quadrivalent Inactivated Vaccine — A seasonal quadrivalent inactivated influenza vaccine (IIV4), prepared from influenza viruses propagated in embryonated chicken eggs, protecting against 2 influenza A subtypes and 2 influenza B subtypes: A/Singapore/GP1908/2015 (H1N1) IVR-180 (an A/Michigan/45/2015 [H1N1] pdm09-like virus), A/Singapore/INFIMH-16-0019/2016 (H3N2) NIB-104, B/Maryland/15/2016 NYMC BX-69A (a B/Colorado/06/2017-like virus), and B/Phuket/3073/2013.

SUMMARY:
The study will be designed as a prospective surveillance of the immune response to seasonal influenza vaccination in 240 healthy children and adults ages 9 and over. Study duration will be 5 years, with a participant duration of 6 months. Subjects will receive a quadrivalent inactivated influenza vaccine, at a dose of not less than 15 ug of hemagglutinin (HA), by intramuscular injection in open label fashion on day 0. Blood draws will occur at baseline, day 7, 28 and 90. The primary objective of this study is to evaluate the relationship between first influenza A virus exposure (inferred by age), vaccine history, and baseline serum antibody response to seasonal influenza vaccine in healthy adults and children.

DETAILED DESCRIPTION:
The study will be designed as a prospective surveillance of the immune response to seasonal influenza vaccination in 240 healthy children and adults ages 9 and over. Study duration will be 5 years, with a participant duration of 6 months. Subjects will receive a quadrivalent inactivated influenza vaccine, at a dose of not less than 15 ug of hemagglutinin (HA), by intramuscular injection in open label fashion on day 0. Blood draws will occur at baseline, day 7, 28 and 90. The primary hypothesis being tested in this study is that there will be differences in the specificity and magnitude of the HA-specific B cell response depending on the age, previous vaccine history and baseline B cell reactivity. The primary objective of this study is to evaluate the relationship between first influenza A virus exposure (inferred by age), vaccine history, and baseline serum antibody response to seasonal influenza vaccine in healthy adults and children. The secondary objective is to evaluate factors related to failure of vaccine to provide protection against symptomatic influenza and the immune response to infection in vaccinated individuals by prospective surveillance of the vaccine cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Aged equal to or greater than 9 years of age and weigh at least 50 pounds
2. The subject must be in good health, as determined by: medical history; and targeted physical examination, when necessary, based on medical history. Stable medical or psychiatric condition is defined as: no recent increase in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months
3. The subject is able to understand and comply with the planned study procedures, including being available for all study visits
4. The subject/parent has provided informed consent/assent prior to any study procedures
5. Subjects who have not received seasonal flu vaccine for the current year

Exclusion Criteria:

1. Subject report of known hypersensitivity to allergy to components of the study vaccine or other components of the study vaccine
2. Subject report of known latex allergy
3. Subject report of a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines
4. Subject report of a history of Guillain-Barre syndrome within 6 weeks of receipt of a previous influenza vaccine
5. The subject is a female of childbearing potential who is currently pregnant or breastfeeding or intends to become pregnant during the study period between enrollment and 90 days following receipt of vaccine. Pregnancy will be determined by subject interview. Pregnancy testing is not done in this study since there is no increased risk in pregnancy
6. The subject is immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months
7. The subject has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years
8. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as per age as using inhaled high dose per reference chart https://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines/quick-reference-html#estimated-comparative-daily-doses
9. The subject received immunoglobulin or another blood product within the 3 months prior to enrollment in this study
10. The subject has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days after vaccination
11. The subject has an acute or chronic medical condition that, in the opinion of the investigator or appropriate sub-investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include any acute or chronic medical disease or conditions defined as persisting for 3 months (defined as 90 days) or longer, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses of the subject's successful completion of the study
12. Subjects with an active infection or that has an acute illness or an oral temperature greater than 99.9 degrees Fahrenheit (37.7 degrees Celsius) within 3 days prior to enrollment or vaccination. Subjects who had an acute illness that was treated symptoms resolved are eligible to enroll as long as treatment is completed and symptoms resolved > 3 days prior to enrollment
13. The subject is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study, or intends to donate blood during the study period
14. The subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
15. The subject has a history of alcohol or drug abuse in the 5 years prior to enrollment
16. The subject has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection
17. Subject weighs less than 50 lbs
18. Subject expects to have a medical procedure during the upcoming 8 weeks that estimates blood loss to exceed 400 cc for adults or for children would exceed 3 ml/kg

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rochester General Hospital - Infectious Disease Unit, Rochester, New York
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults and children ages 9 and over
Period: Overall Study
Arm/Group | Arm 1
Started | 152
Completed | 141
Not Completed | 11
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Early Study Termination due to COVID-19 pandemic | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 109
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 43 [9 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 139
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 137
  More than one race | 4
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Magnitude of the Serum Antibody Response by Hemagglutination-inhibition (HAI)
Description: A/Hong Kong/4801/2014 (H3N2) day 28 Season 2017-2018
Time Frame: Through Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | Arm 1
Number analyzed (Participants) | 18
titer | 528 (1.38)

2. Primary Outcome: Magnitude of the Serum Antibody Response by Microneutralization (MN)
Description: A/Hong Kong/4801/2014 (H3N2) Day 28 MN Season 2017-2018
Time Frame: Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | Arm 1
Number analyzed (Participants) | 18
titer | 806 (1.21)

3. Primary Outcome: Serum Antibody Response by Hemagglutination-inhibition (HAI)
Description: A/Hong Kong/4801/2014 (H3N2) Day 90 Season 2017-2018
Time Frame: Day 90
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | Arm 1
Number analyzed (Participants) | 17
titer | 115 (3.08)

4. Primary Outcome: Serum Antibody Response by Microneutralization (MN)
Description: A/Hong Kong/4801/2014 (H3N2) Day 90 MN Season 2017-2018
Time Frame: Day 90
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | Arm 1
Number analyzed (Participants) | 17
titer | 1389 (1.08)

5. Primary Outcome: Specificity of the Serum Antibody Response by Hemagglutination-inhibition (HAI)
Description: A/H1N1/Michigan/45/2015 pdm09 Day 28 Season 2017-2018
Time Frame: Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | Arm 1
Number analyzed (Participants) | 18
titer | 665 (1.73)

6. Primary Outcome: Specificity of the Serum Antibody Response by Microneutralization (MN)
Description: A/H1N1/Michigan/45/2015 pdm09 Day 28 Season 2017-18
Time Frame: Day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: titer
Arm/Group | Arm 1
Number analyzed (Participants) | 18
titer | 2281 (2.86)

7. Secondary Outcome: Age at Time of First Influenza A Exposure
Description: Comparison between groups: subjects who develop symptomatic influenza (Vaccine Failures) vs. subjects who do not
Time Frame: Baseline
Reporting Status: Not Posted

8. Secondary Outcome: Baseline B Cell Reactivity
Description: Comparison between groups: subjects who develop symptomatic influenza (Vaccine Failures) vs. subjects who do not
Time Frame: Baseline
Reporting Status: Not Posted

9. Secondary Outcome: Vaccine History (Number and Percentage of Participants to Receive Vaccine)
Description: Comparison between groups: subjects who develop symptomatic influenza (Vaccine Failures) vs. subjects who do not
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/152
Serious Adverse Events (participants affected / at risk) | 1/152
Other Adverse Events (participants affected / at risk) | 24/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=152)
Gastric Mass, S/P Wedge resection, GIST Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=152)
Upper Respiratory Tract Infection (Infections and infestations) | 24 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT03328325/Prot_SAP_000.pdf